CLINICAL TRIAL: NCT04626141
Title: Time to Healing, Loss of Fixation, and Loss of Alignment in Supracondylar Distal Femur Fractures Among a Geriatric Population Treated With Abaloparatide: A Double-Blind Placebo Controlled Study
Brief Title: Supracondylar Distal Femur Fractures and Abaloparatide
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn due to staffing/enrollment related challenges.
Sponsor: Daniel Horwitz (Other)
Collaborators: Radius Health, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Horwitz, Principal Investigator, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0544
Record Dates: First submitted 2020-09-30; First posted 2020-11-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures | interventions — abaloparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abaloparatide group (Experimental): Patients in the experimental group will receive abaloparatide after their surgery.
  Interventions: Drug: Abaloparatide
- Control group (Placebo Comparator): Patients in the control group will receive a placebo after their surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abaloparatide — Abaloparatide will be dispensed as a 30-day supply of disposable pen injections of the standard, FDA approved dosage (80 mcg abaloparatide).
  Arms: Abaloparatide group
Drug: Placebo — Placebo will be dispensed as a 30-day supply of disposable pen injections.
  Arms: Control group

SUMMARY:
Supracondylar femur fractures in the geriatric population present a unique challenge to the orthopaedic surgeon both in terms of fixation, healing, and final extremity axial alignment. Pulsed dosing of parathyroid hormone derivatives (Forteo) has been shown to increase bone mass, and several studies in Europe have demonstrated its benefit as an adjuvant for fracture healing. Abaloparatide represents a new compound which similarly offers great potential for accelerating fracture healing, especially healing associated with callous formation. This is a randomized, double blind placebo-controlled trial to compare a group of patients being treated for supracondylar distal femur fractures who receive abaloparatide (n=38) with a control group of patients who receive a placebo (n=38).

DETAILED DESCRIPTION:
Supracondylar femur fractures in the geriatric population present a unique challenge to the orthopaedic surgeon both in terms of fixation, healing, and final extremity axial alignment. Multiple methods of fixation are well accepted, and each has its own advantages and disadvantages. The common occurrence of periprosthetic supracondylar femur fractures adds another level of complexity, and the universal goal when treating these patients is to obtain and maintain acceptable alignment, allow mobilization and early weight bearing, and achieve union. To a degree, mobilization and weight bearing compete with maintenance of axial alignment, and any final outcome is a race between healing and loss of fixation. As a result, any intervention that can accelerate healing would be of great benefit. As the vast majority of these injuries heal with secondary bone healing (callous), the determination of "healing" is reliably determined using the modified Radiographic Union Score for Tibia Fractures (mRUST), and thus this patient population offers an ideal population in which to evaluate an accelerant of fracture healing.

Pulsed dosing of parathyroid hormone derivatives (Forteo) has been shown to increase bone mass, and several studies in Europe have demonstrated its benefit as an adjuvant for fracture healing. Abaloparatide represents a new compound which similarly offers great potential for accelerating fracture healing, especially healing associated with callous formation. This is a randomized, double blind placebo-controlled trial to compare a group of patients being treated for supracondylar distal femur fractures who receive abaloparatide (n=38) with a control group of patients who receive a placebo (n=38).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 65 years old
2. Subject is willing and able to read, comprehend, and sign the study informed consent form in English prior to study specific procedure
3. Subject is being treated for a closed supracondylar distal femur fracture with either a retrograde nail or locked plate
4. Subject undergoes open reduction/fixation

Exclusion Criteria:

1. Subject has open fracture
2. Bilateral injury or other lower extremity injury that would affect weight bearing status
3. Subject's postoperative radiographs (on day of surgery) indicate failure to achieve axial alignment (more than 10 degrees axial alignment and more than 25% anterior/posterior displacement in lateral view)
4. Subject has additional severe traumatic conditions such as closed head injury
5. Subject has medical condition or is on medication that may significantly affect healing (i.e. immunosuppressive diseases and drugs)
6. Subject has active or history of Paget's disease of the bone, bone cancer, or other bone diseases or conditions placing them at increased risk of osteosarcoma
7. Subject has active or history of hypercalcemia or underlying hypercalcemic disorder, such as primary hyperparathyroidism
8. Subject has active or a history of urolithiasis
9. Subject will have trouble injecting the pen and does not have someone to help them on a daily basis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
modified Radiographic Union Score for Tibia Fractures (mRUST) | 6 weeks
  degree of callous formation and healing (worst 4 - 16 best)
maintenance of axial alignment and loss of fixation | 6 weeks
  change in the angle between the surface and fixed implant from the baseline radiographs (taken immediately postoperative) and the radiographs taken at 6, 12, and 24 weeks postoperative

SECONDARY OUTCOMES:
modified Radiographic Union Score for Tibia Fractures (mRUST) | 12 weeks
  degree of callous formation and healing (worst 4 - 16 best)
modified Radiographic Union Score for Tibia Fractures (mRUST) | 24 weeks
  degree of callous formation and healing (worst 4 - 16 best)
maintenance of axial alignment and loss of fixation | 12 weeks
  change in the angle between the surface and fixed implant from the baseline radiographs
maintenance of axial alignment and loss of fixation | 24 weeks
  change in the angle between the surface and fixed implant from the baseline radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Horwitz, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States